CLINICAL TRIAL: NCT03112798
Title: Miller vs Macintosh Size 0 Blades for Tracheal Intubation of Infants Under 1 Month: a Randomized Comparative Study
Brief Title: Miller vs Macintosh Size 0 Blades for Tracheal Intubation of Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Science University (Other)
Responsible Party: Principal Investigator, Kemal Tolga Saracoglu, Associate Professor MD, Istanbul Science University
Other Study IDs: 44140529/2016-50
Record Dates: First submitted 2017-03-23; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Newborn
Keywords: tracheal intubation; Macintosh blade; Miller blade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Macintosh group: The patients will be intubated by using Macintosh blades and the outcomes will be compared with Miller blades.
- Miller group: The patients will be intubated by using Miller blades and the outcomes will be compared with Macintosh blades.

SUMMARY:
Miller blades are commonly used in pediatric anesthesia; however, there is less evidence-based information on the superiority of Miller blades in the visualization of the laryngeal inlet to Macintosh blades. The aim of the present study is to compare the glottic views with the size 0 Macintosh and Miller laryngoscope blades above and below the epiglottis.

DETAILED DESCRIPTION:
Miller blades are commonly used in pediatric anesthesia; however, there is less evidence-based information on the superiority of Miller blades in the visualization of the laryngeal inlet to Macintosh blades (1,2). Therefore prospective randomized comparative studies on this field is required. Passi et al. (3) have demonstrated that, in 50 children aged between 6 months and 2 years, optimal laryngeal views could be obtained with either the Miller size 1 blades lifting the epiglottis or with Macintosh size 1 blades lifting the tongue base. Another clinical trial compared the laryngoscopic views and tracheal intubation conditions with Macintosh and Miller blades in children from 1 month to 24 months. In this study involving 120 children, similar glottic views were obtained with both blades in 43% of the children while a better view was observed with the Miller blade in 29% of the children and with the Macintosh blade in 28% (4). Direct laryngoscopy for tracheal intubation in neonates is a procedure that mostly requires experience and constant practice (5). Neonates have a number of distinctive airway characteristics. These characteristics include the large tongue and head, the floppy, narrow U-shaped epiglottis, the larynx that is located more cephalad, and the vocal cords that are angled in an anterior-caudal position (4). Therefore, straight laryngoscope blades are recommended for use in children and infants under 2 years of age.

In neonatal tracheal intubations, Miller blade is the most frequently utilized blade (6). The reasons for this include the effective displacement of the tongue to the left of the laryngoscope with the Miller blade and the effective lifting of the long and floppy epiglottis during laryngoscopy (3). However, there is no prospective randomized and blinded comparative clinical study on this subject. The aim of the present study is to compare the glottic views with the size 0 Macintosh and Miller laryngoscope blades above and below the epiglottis.

Methods:

For the present study, the Ethics Committee approval was be obtained from the Faculty of Medicine, Istanbul Science University. Written informed consent will be obtained from the parents of patients undergoing elective surgery. The study will involve ASA I or II patients under 1 month. Infants with a history of a difficult airway or diagnosed congenital syndrome, premature infants less than 37 weeks gestational age at birth, and those with acute or chronic pulmonary or neuromuscular diseases will be excluded from the study. Twenty five children undergoing elective surgery will be enrolled in the study. Infants will be randomized (using www.random.com) into two groups, the Miller and Macintosh blade groups, and whether the assigned blade is inserted above or below the epiglottis first, with allocation stored within sealed opaque envelopes until consent is obtained.

In a standard monitoring process, electrocardiogram (ECG), oxygen saturation, non-invasive blood pressure (NIBP), temperature and end-tidal CO2 pressure (EtCO2) will be monitored. Following the monitoring, anesthesia will be induced with 50% air, 50% oxygen and 8% sevoflurane. Once intravenous access is obtained, 0.5 mg/kg rocuronium will be administered. After preoxygenating with 100% oxygen and sevoflurane for 3 minutes, the assigned blade will be inserted into the mouth. All laryngoscopies will be performed by one of three paediatric anesthetists. The Miller blade will be inserted into the mouth at the right commissure and the tongue swept gently to the left. The best laryngeal view will be achieved by optimizing the head position and applying external pressure to the larynx. As described by Passi et al. (3), two laryngeal views will be obtained with the same blade in each patient: lifting the epiglottis or the tongue base. The order of the views (lifting the epiglottis or the tongue base) will be determined by randomization immediately before laryngoscopy. The laryngeal views will be photographed each time by an anesthetist using a digital Olympus camera without using flash. The camera will be optimally positioned before laryngoscopy in order to capture the best possible views. The photos will be reviewed by a blinded anesthetist using the percentage of glottic opening (POGO) score (7,8). This anesthetist will be blinded to the study hypothesis as well as which blade was used and where it was placed. We will photo the child's name and the randomization code-blade type and which view was taken before and after each photo of the larynx. Then the photos will be uploaded and the number of the photo will be recorded in the study record for the child so we will know which photo corresponds to which blade and position for each child. After all the photos are taken, they will be randomized and given to the blinded observer to measure the vocal cord span.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II patients under 1 month.

Exclusion Criteria:

* Infants with a history of a difficult airway or diagnosed congenital syndrome, premature infants less than 37 weeks gestational age at birth, and those with acute or chronic pulmonary or neuromuscular diseases will be excluded from the study.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include newborns
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
POGO scores | five months
  the laryngeal views will be photographed during laryngoscopy and will be compared

SECONDARY OUTCOMES:
complications | five months
  any complication will be recorded during tracheal intubation with each device

CONTACTS AND LOCATIONS:
Overall Officials: Kemal T Saracoglu, Principal Investigator — Istanbul Science University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] DAVENPORT HT, ROSALES JK. Endotracheal intubation of infants and children. Can Anaesth Soc J. 1959 Jan;6(1):65-74. doi: 10.1007/BF03014197. No abstract available. PMID 13608313
- [Result] Jones RM, Jones PL, Gildersleve CD, Hall JE, Harding LJ, Chawathe MS. The Cardiff paediatric laryngoscope blade: a comparison with the Miller size 1 and Macintosh size 2 laryngoscope blades. Anaesthesia. 2004 Oct;59(10):1016-9. doi: 10.1111/j.1365-2044.2004.03839.x. PMID 15488063
- [Result] Passi Y, Sathyamoorthy M, Lerman J, Heard C, Marino M. Comparison of the laryngoscopy views with the size 1 Miller and Macintosh laryngoscope blades lifting the epiglottis or the base of the tongue in infants and children <2 yr of age. Br J Anaesth. 2014 Nov;113(5):869-74. doi: 10.1093/bja/aeu228. Epub 2014 Jul 25. PMID 25062740
- [Result] Varghese E, Kundu R. Does the Miller blade truly provide a better laryngoscopic view and intubating conditions than the Macintosh blade in small children? Paediatr Anaesth. 2014 Aug;24(8):825-9. doi: 10.1111/pan.12394. Epub 2014 Apr 2. PMID 24690084
- [Result] Lingappan K, Arnold JL, Shaw TL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2015 Feb 18;(2):CD009975. doi: 10.1002/14651858.CD009975.pub2. PMID 25691129
- [Result] Fiadjoe JE, Gurnaney H, Dalesio N, Sussman E, Zhao H, Zhang X, Stricker PA. A prospective randomized equivalence trial of the GlideScope Cobalt(R) video laryngoscope to traditional direct laryngoscopy in neonates and infants. Anesthesiology. 2012 Mar;116(3):622-8. doi: 10.1097/ALN.0b013e318246ea4d. PMID 22270505
- [Result] Levitan RM, Ochroch EA, Kush S, Shofer FS, Hollander JE. Assessment of airway visualization: validation of the percentage of glottic opening (POGO) scale. Acad Emerg Med. 1998 Sep;5(9):919-23. doi: 10.1111/j.1553-2712.1998.tb02823.x. PMID 9754506
- [Result] Ochroch EA, Hollander JE, Kush S, Shofer FS, Levitan RM. Assessment of laryngeal view: percentage of glottic opening score vs Cormack and Lehane grading. Can J Anaesth. 1999 Oct;46(10):987-90. doi: 10.1007/BF03013137. PMID 10522589